CLINICAL TRIAL: NCT02655783
Title: Utilisation parentérale de Normal Salin Avec ou Sans Dextrose Durant l'Induction du Travail Chez Les Nullipares
Brief Title: Use of Normal Saline With or Without Dextrose During Induction of Labor in Nulliparous
Acronym: DEXTRONS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 12-143
Record Dates: First submitted 2015-03-04; First posted 2016-01-14 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Delivery Uterine
Keywords: induction of labor
MeSH Terms: interventions — Glucose; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Active Comparator): normal saline, 250 ml/h, until expulsion of placental
  Interventions: Other: normal saline
- intervention (Experimental): normal saline + 5% dextrose, 250 ml/h, until expulsion of placental
  Interventions: Other: 5% dextrose; Other: normal saline

INTERVENTIONS:
Other: 5% dextrose — women with an elective induction of labor receive IV hydratation (250 ml/h) with a normal saline solution + 5% dextrose
  Arms: intervention
Other: normal saline — women with an elective induction of labor receive IV hydratation (250 ml/h) with a normal saline solution

SUMMARY:
The objective of this study is to compare the effects of use of normal saline (250 cc / h), with or without dextrose supplement, on the evolution of labor in nulliparous.

DETAILED DESCRIPTION:
There is some controversy regarding intravenous hydration of patients during labor. While the use of a fast flow of hydration appears to be recognized beneficial, the addition of glucose is less well accepted. However studies on exercise physiology clearly demonstrates improved performance of skeletal muscle by increased hydration and carbohydrate replacement during prolonged exercise. This situation is similar to the condition of the uterus in labor especially since it is now established that glucose represents its principal source of energy.

However, the effect of an additional carbohydrate intake on the evolution of labor has not been extensively studied until now, and there are several schools of thought on this subject. While some studies show that such glucose addition could reduce the total duration of labor as well as its second stage, others claim that this glucose supplement offers no benefit and may even be harmful to the fetus.

It therefore seems imperative to conduct a study to compare the use of hydration with normal saline with or without dextrose during labor, as recommended in current flow (250 cc / h). To our knowledge, this has never been done.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous woman
* monofetal pregnancy
* delivery at term
* elective induction
* favorable cervix (Bishop score of at least 6)
* cephalic presentation

Exclusion Criteria:

* diabetes
* preeclampsia
* maternal heart disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-01; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
2nd stage of labor | during delivery of a first baby, for an average of 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yves-André Bureau, MD, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Oral presentation at the Society of Maternal and Fetal Medicine annual meeting (January 2017, Las Vegas) Manuscript in preparation